CLINICAL TRIAL: NCT06098456
Title: Treatment With Epigallcoatechin Gallate, Hyaluronic Acid, Folic Acid and Vitamin B12 in Women HPV Positive With Abnormal Cytology Tests
Brief Title: Epigallocatechin Gallate and Other Antural Compounds in HPV Infections
Acronym: EGCGHPV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro di Ricerca Clinica Salentino (Network)
Responsible Party: Principal Investigator, ANDREA TINELLI, Professor, Centro di Ricerca Clinica Salentino
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPV-EGCG
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Papilloma-induced Cervical Lesions
Keywords: EGCG; HPV; Folic acid; Hyaluronic acid; Vitamin B12; LSIL
MeSH Terms: interventions — epigallocatechin gallate; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: Patients decide wheter to receive the experimental treatment or to undergo routine clinical practice.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): The patients in this group undergo treatment with Epigallocatechin gallate 200mg, Hyaluronic acid 50mg, Vitamin B12 1mg and Folic acid 400mcg by oral route once per day.
  Interventions: Drug: EGCG, FA, HA, B12
- Control (No Intervention): The patients in this group follow the routine clinical practice, namely the clinical monitoring.

INTERVENTIONS:
Drug: EGCG, FA, HA, B12 — Epigallocatechin gallate 200mg, Hyaluronic acid 50mg, Vitamin B12 1mg, Folic acid 400mcg
  Other Names: Pervistop
  Arms: Treatment

SUMMARY:
The investigators enroll patients with a PAP-test cytology reporting LSIL or ASCUS.

Pateitns undergo HPV-DNA test for screening. Patients are treated with Epigallocatechin galalte, hyaluronic acid, folic acid and Vitamin B12 by oral route.

After three months of treatment PAP-test and HPV-DNA test will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Positivity to HPV-DNA test
* PAP-test reporting LSIL or ASCUS

Exclusion Criteria:

* HPV-related pathologies or complicances apart from LSIL or ASCUS
* Diagnosis of cancer

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Positivity to HPV infection | 3 and 6 months
  The outcome consists of the number of negative DNA-test obtained in patients previously positive.

SECONDARY OUTCOMES:
Occurrence of lesions | 3 and 6 months
  The outcome consists of the number of negative PAP-tests obtained in patients previously positive.
Lesions-related symptmos | 3 and 6 months
  The ouctome includes the occurrence of bleeding, flogosis, or sexual pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Veris delli Ponti, Scorrano, Lecce, Italy